CLINICAL TRIAL: NCT04809155
Title: A Reproductive Health Program for A Select Population
Brief Title: Girl2Girl: A Web-based Trial
Acronym: G2G
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Center for Innovative Public Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01HD095648 (NIH)
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Pregnancy Prevention
Keywords: Teenage Pregnancy Prevention; LGB Girls; Text messaging

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Girl2Girl (Experimental): Girls receive text messages that address the information, motivation, and behavioral skills components need to prevent unwanted pregnancy.
  Interventions: Behavioral: Girl2Girl
- Control - Healthy lifestyle (No Intervention): Girls receive text messages about a 'healthy lifestyle', including healthy social media use and self-esteem.

INTERVENTIONS:
Behavioral: Girl2Girl — The program has a 'core' 7 weeks of daily messages and then a week 'booster' that is delivered 3 months later.
  Arms: Girl2Girl

SUMMARY:
This is a pilot effectiveness study of Girl2Girl, a text messaging-based pregnancy prevention program for cisgender sexual minority adolescents.

DETAILED DESCRIPTION:
An estimated one in four teen women will become pregnant by the time she is 20 years of age. That said, significant disparity in rates exist for lesbian, gay, bisexual and other sexual minority women (LGB) versus non-LGB teen women: Research suggests that lesbian and bisexual teen women are between two and four times more likely to report having been pregnant than teen women who identified as exclusively heterosexual. Despite this compelling evidence that lesbian and bisexual adolescent women are at risk for teen pregnancy, programs tailored to the unique needs of adolescent LGB women are nonexistent. Evidence-based teen pregnancy prevention (TPP) programs targeting LGB teen women are urgently needed.

The Girl2Girl intervention text messaging-based TPP program designed specifically for LGB women ages 14-18 years, nation-wide. This is an extension of a previous randomized controlled trial. Here, the cohort was recruited using an effectiveness strategy: Girls were allowed to register and enroll themselves without needing to talk to research staff. All eligible and interested youth were allowed to enroll; no diversity targets were applied.

ELIGIBILITY:
Inclusion Criteria:

* Endorse a non-heterosexual sexual identity (i.e., lesbian/gay, bisexual, queer, questioning, unsure) on the screener;
* Be cisgender (i.e., be assigned a female sex at birth and endorse a female gender identity) on the screener;
* Be aged 14-18;
* Be English speaking;
* Be able to provide informed assent, including the self-directed self-safety assessment.

Exclusion Criteria:

* Not passing the self-directed self-safety assessment
* Knowing someone who is already enrolled in the program (added part-way through the recruitment period)
* Non-cisgender identity in the screener

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Youth self-identified as cisgender female in the screener.
Enrollment: 574 (Estimated)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-06-07 (Estimated); Study Completion 2021-06-07 (Estimated)

PRIMARY OUTCOMES:
Number of Condom protected penile-vaginal Sex Acts | 3-months post-intervention
  The relative difference of protected penile-vaginal sex acts in the intervention versus control group at 3-months post-intervention
Number of Participants Who Used Other Birth Control Methods | 3-months post-intervention
  The relative difference of teens who used birth control methods other than condoms (e.g., the pill, the patch) in the intervention versus control group at 3-months post-intervention

SECONDARY OUTCOMES:
Testing for HIV and other sexually transmitted infections (STIs) | 3-months post intervention
  The relative odds of reporting an HIV or other STI test during the observation period for those in the intervention versus control
Pregnancy | 3-months post intervention
  The percent of teens who have been pregnant since the beginning of the observation period in the intervention versus control group
Intentions to use condoms | 3-months post intervention
  The percent of teens who intend to use condoms if they have penile-vaginal sex in the future
Intentions to Use Birth Control Other Than Condoms | 3-months post intervention
  The percent of teens who intend to use birth control other than condoms if they have penile-vaginal sex in the future

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Innovative Public Health Research, San Clemente, California, United States

IPD SHARING:
Plan to Share IPD: No